CLINICAL TRIAL: NCT07268911
Title: Femoral Rami Obturator Nerve Trunk (FRONT) Block in Intramedullary Nail Surgery .
Acronym: FRONT block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gaber Ahmed, lecturer in anesthesia, Intensive Care and Pain Management, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ِAIP029-4
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Anterior Hip Analgesia
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block Group (Active Comparator): will receive FRONT block
  Interventions: Procedure: Femoral rami obturator nerve trunk (FRONT) block
- Control group (No Intervention): will receive conventional analgesia

INTERVENTIONS:
Procedure: Femoral rami obturator nerve trunk (FRONT) block — ultrasound-guided FRONT block will be performed at the infrainguinal level, targeting the iliopsoas plane. Using the same needle approach, the subpectineal compartment will be also accessed . We will use ultrasound and electrical nerve stimulation guidance (0.4 mA, 0.1 ms, without eliciting a motor response) to avoid direct involvement of the femoral nerve. A total of 40 mL (20 mL for the iliopsoas plane and 20 mL for the subpectineal compartment) of 0.125% plain levobupivacaine will be administered.
  Arms: Block Group

SUMMARY:
The study propose that using femoral rami obturator nerve trunk(FRONT) block may help postoperative analgesia in nail femur surgeries. The technique is relatively new, introducing one needle to target two nerve blocks in the same entry point. The block spare motor fibers of femoral nerve so it may help both early mobilization and effective analgesia, which in turn enhance early recovery and better outcomes.

DETAILED DESCRIPTION:
Post operative pain levels after hip fracture are high during ambulation and may worsen outcome after hip fracture. Regional anesthesia has shown to facilitate rehabilitation in orthopedics procedures. Many of these regional anesthesia techniques ,such as femoral nerve, lumber plexus, peri capsular nerve group(PENG), fascia iliaca blocks have gained attention for their opioid and some times for motor sparing potential, as well as the ability to provide targeted analgesia for anterior hip joint. Nevertheless the anterior hip joint coverage needs the constant contribution of femoral and obturator nerves to provide adequate pain relieve. In this study patients will receive preoperative femoral rami obturator nerve trunk(FRONT) block , a novel regional anesthesia technique described by Jessen et al., as a promising solution to the long-standing challenge of anesthetizing both the femoral and obturator nerve branches in anterior hip joint for postoperative pain control, addressing a more comprehensive coverage of anterior hip innervation.

ELIGIBILITY:
Inclusion Criteria:

* the elderly age≥60 years
* American Society of Anesthesiologists (ASA) classification 1-2
* patients who undergoing surgery for intramedullary nail surgery.

Exclusion Criteria:

* patient refused to participate and consent
* patients with a history of mild cognitive impairment (MCI), dementia, and delirium
* patients with known preoperative infections (pulmonary infection, urinary infection, and sepsis).
* coagulopathy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesia | Patients will be followed for 36 hours postoperatively and assessed for pain, at 2, 4, 6, 12, 18, 24, 36 hours
  Pain level will be assessed after spinal anesthesia is resolved using rest/dynamic numeric rating scale (NRS) with patients rating their pain on a scale from 0 to 10. On this scale, 0 means "no pain" and 10 means "the worst pain imaginable"

SECONDARY OUTCOMES:
Opioid consumption | When 36 hours postoperatively has passed.
  First analgesic request time and total opioid consumption will be recorded
Motor function | Patients will be followed for 36 hours postoperatively and assessed for motor function at 2, 4, 6, 12, 18, 24, 36 hours.
  Motor function will be assessed using Modified Bromage scale after spinal anesthesia has been resolved, where score 0 means full movement, and 4 means complete motor loss.
Complication | Patients will be followed for 36 hours postoperatively and assessed for presence of any complications or side effects at 2, 4, 6, 12, 18, 24, 36 hours
  any complication either surgical or side effects will be recorded (vomiting, allergy, urinary retention, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab M Sayed, MD, Study Director — Qena University
Locations (1):
- Qena University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No